CLINICAL TRIAL: NCT02366494
Title: Utility of Exosomal MicroRNAs to Predict Response to Androgen Deprivation Therapy in Prostate Cancer Patients
Brief Title: Micro RNAs to Predict Response to Androgen Deprivation Therapy
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Deepak Kilari, Associate Professor, Medical College of Wisconsin
Other Study IDs: 23842
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; treatment response; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Leuprolide; Goserelin; Triptorelin Pamoate; Docetaxel; abiraterone; Abiraterone Acetate; apalutamide; enzalutamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood collection at pre treatment (at enrollment), 3 months post treatment, and at the time of disease progression (or at 2 years post treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Androgen blockade: Androgen DeprivationTherapy or Complete Androgen Blockade
  Interventions: Drug: Bicalutamide; Drug: Leuprolide; Drug: Goserelin; Drug: Triptorelin
- Hormonal Therapy and Chemotherapy: Hormonal therapy, novel oral hormonal therapy (abiraterone/apalutamide/enzalutamide) and chemotherapy (docetaxel)
  Interventions: Drug: Bicalutamide; Drug: Leuprolide; Drug: Goserelin; Drug: Triptorelin; Drug: Docetaxel; Drug: Abiraterone; Drug: Apalutamide; Drug: Enzalutamide

INTERVENTIONS:
Drug: Bicalutamide — ANDROGEN BLOCKADE
  Other Names: Casodex
Drug: Leuprolide — ANDROGEN BLOCKADE
  Other Names: Lupron
Drug: Goserelin — ANDROGEN BLOCKADE
  Other Names: Zoladex
Drug: Triptorelin — ANDROGEN BLOCKADE
  Other Names: Trelstar
Drug: Docetaxel — Chemo hormonal therapy
  Other Names: Taxotere
  Groups: Hormonal Therapy and Chemotherapy
Drug: Abiraterone — Chemo hormonal therapy
  Other Names: Zytiga
  Groups: Hormonal Therapy and Chemotherapy
Drug: Apalutamide — Nonsteroidal antiandrogen medication
  Other Names: Erleada
  Groups: Hormonal Therapy and Chemotherapy
Drug: Enzalutamide — Nonsteroidal antiandrogen medication
  Other Names: Xtandi
  Groups: Hormonal Therapy and Chemotherapy

SUMMARY:
Identify exosomal micro RNA that predict responses to ADT

DETAILED DESCRIPTION:
1. Identify novel exosomal RNA signatures at pretreatment that predict response to ADT.

   The study team will collect blood samples from patients with systemic disease pretreatment (at enrollment), three months post-treatment and at the time of progression of disease (or at two years post-ADT for patients still in remission at that time point) and then perform next-generation sequencing using serum exosomal RNAs derived from these patients.

   The investigators plan to identify exosomal RNAs signatures that change between pretreatment (at enrollment) and during treatment (at three months) and further explore the effect of these changes on disease response. The investigators also plan to compare exosomal RNA levels between patients relapse within the first two years versus those in remission at two years. Among patients with progression, the investigators plan to compare exosomal RNA signatures at progression of disease to signatures at pretreatment and during treatment.
2. Validate exosomal RNA markers that predict response to ADT by real-time RT-PCR.

Secondary objectives: Selected RNAs, identified through the above process will be validated using real-time RT-PCR assay to test reproducibility of RNA sequencing results. The investigators expect to select and validate approximate five RNA markers that predict duration of response to ADT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer.
* Testosterone level >30ng/ml and at least 6 months since last dose of hormonal therapy.
* History/physical examination including a detailed description of the stage of prostate cancer within 8 weeks prior to registration.
* CT scan of abdomen and pelvis with IV contrast and bone scan should be performed within 8 weeks prior to registration.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Age ≥ 18.
* Patients must provide study-specific informed consent prior to study entry for this project and mandatory blood specimen for banking for future studies (future studies may include genetic testing).

Exclusion Criteria:

* Received hormonal therapy less than 6 months prior to registration.
* History of active secondary malignancy.
* Decline hormone therapy for prostate cancer.
* Current or previous treatment with 5-alpha reductase inhibitors within 6 months prior to enrollment.

Ages: 21 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with systemic disease ( with biochemical relpase or metastaic disease)
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Identify five most prevalent exosomal microRNAs that predict response to androgen deprivation therapy based treatment. | Up to two years
  Two hundred to 300 microRNAs will be identified by RNA sequencing. This outcome measure will report the read count per million of the top-five most prevalent microRNAs that correlate with responses.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kilari, MD, Principal Investigator — The Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Huggins C, Hodges CV. Studies on prostatic cancer. I. The effect of castration, of estrogen and androgen injection on serum phosphatases in metastatic carcinoma of the prostate. CA Cancer J Clin. 1972 Jul-Aug;22(4):232-40. doi: 10.3322/canjclin.22.4.232. No abstract available. PMID 4625049
- [Background] Taplin ME, Xie W, Bubley GJ, Ernstoff MS, Walsh W, Morganstern DE, Regan MM. Docetaxel, estramustine, and 15-month androgen deprivation for men with prostate-specific antigen progression after definitive local therapy for prostate cancer. J Clin Oncol. 2006 Dec 1;24(34):5408-13. doi: 10.1200/JCO.2006.06.6589. PMID 17135641